CLINICAL TRIAL: NCT01468116
Title: The Effect of Roux-en-Y Gastric Bypass on Mitochondrial Function in Type 2 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Anna Kirstine Bojsen-Moeller, MD, Hvidovre University Hospital
Other Study IDs: MITBypass
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Type 2 diabetes; Gastric bypass surgery; Obesity; Mitochondrial function
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- RYGB patients with type 2 diabetes: Morbidly obese patients with type 2 diabetes undergoing gastric bypass surgery
- RYGB patients without type 2 diabetes: Morbidly obese patients with normal glucose tolerance undergoing gastric bypass surgery
- Cholecystectomy patients without type 2 diabetes: Patients with normal glucose tolerance undergoing laparoscopically cholecystectomy

SUMMARY:
Roux-en-Y gastric bypass (RYGB) surgery induces resolution of type 2 diabetes, often within days after surgery and before significant weight loss. The aim of this study is to investigate whether changes in mitochondrial function contributes to the early improvement of type 2 diabetes after RYGB.

DETAILED DESCRIPTION:
Mitochondrial dysfunction has been linked to development of insulin resistance in the muscle and hence to the pathogenesis of type 2 diabetes. Mitochondrial function can be studied non-invasively by 31 Phosphor Magnetic Resonance spectroscopy (31PMRS). In this study we will investigate changes in mitochondrial function using the combination of 31 PMRS and Near Infra-Red Spectroscopy (NIRS) after gastric bypass.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for gastric bypass surgery or cholecystectomy
* Verified type 2 diabetes or normal glucose tolerance by OGTT

Exclusion Criteria:

* Patients unable to fit the dimensions of the MRI-scanner

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects are recruited from the outpatient clinic of endocrinology and the gastrosurgical clinic at Hvidovre University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-06 (Estimated); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Copenhagen, Hvidovre, Denmark